CLINICAL TRIAL: NCT06465485
Title: STEP: A Prospective, Interventional, Multicenter, Single-Arm Phase 3b Study to Evaluate the Step-Down of Maintenance Therapy in Patients With Severe Eosinophilic Asthma Treated With Benralizumab
Brief Title: STEP: Phase IIIb Study of Benralizumab to Step-down Maintenance Therapy in Patients With Severe Eosinophilic Asthma
Acronym: STEP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3250L00046
Record Dates: First submitted 2024-02-01; First posted 2024-06-18 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benralizumab (Experimental): Severe eosinophilic asthma taking medium-high dose ICS/LABA with/without LTRAs, LAMAs will be all treated by study Drug.
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — Severe eosinophilic asthma taking medium-high dose ICS/LABA with/without LTRAs, LAMAs will be enrolled into this single arm treatment.
  Other Names: Fasenra

SUMMARY:
This is a prospective, multi-center, single-arm Phase 3b study designed to evaluate the potential benefit to patients if benralizumab treatment could enable reduction in asthma maintenance controllers while allowing patients to maintain asthma control in Chinese patients.

DETAILED DESCRIPTION:
The study population will be approximately 480 patients on MD/HD ICS/LABA with and without LTRA or LAMA or theophylline and meeting study inclusion and exclusion criteria in China. After patients sign the informed consent, they will undergo a screening visit (Visit 1, Week -1 to Week 0) to assess eligibility criteria. Patients who meet eligibility criteria and complete study baseline assessments will enter the study and receive the first dose of benralizumab at visit 2 (Week 0).

The benralizumab treatment includes 4 phases: Induction Phase (16 weeks), Reduction Phase (24 weeks), Maintenance Phase (16 weeks) and Follow-up Phase (4 weeks). After initiation of benralizumab 30 mg administered subcutaneously every 4 weeks (Q4W) for the first 3 doses (Visits 2 to 4), then every 8 weeks (Q8W) thereafter.

ELIGIBILITY:
Informed Consent

1．Provision of informed consent prior to any study-specific procedures. Written informed consent, and assent when applicable for study participation must be obtained prior to any study related procedures being performed (local regulations are to be followed in determining the assent/consent requirements for children and parent[s]/guardian[s]) and according to international guidelines and/or applicable local guidelines.

Age 2. Patient must be aged 12-75 years old, inclusively, at the time of Visit 1(Week -1 to Week 0) For those patients, who are 17 on the day of Visit 1(Week -1 to Week 0) but will turn 18 after this day, will be considered an adolescent for the purposes of this study.

Type of Patient and Disease Characteristics 3. Documented history of physician-diagnosed asthma prior to Visit 1

* Documented post-bronchodilator (post-BD) reversibility in FEV1 of ≥12% and ≥200 mL in FEV1 or positive result of branchial provocation test within 12 months prior to Visit 1. If historical documentation is not available, reversibility must be demonstrated and documented at Visit 1.
* Prior to screening (Visit 1, Week -1 to Week 0), patients must have either a documented asthma diagnosis for >6 months or a history of ICS/LABA use for >6 months.

  4. Documented diagnosis of severe eosinophilic asthma (EOS≥150 cells/μL at enrollment, and if EOS 150-<300 cells/μL at enrollment, must have EOS≥300 cells/μL at sometime within 1 year before enrollment) 5. Documented current maintenance treatment with MD/HD ICS + LABA with up to one additional controller
* Other acceptable asthma controller includes LTRA and LAMA 6. On stable MD/HD ICS(>250μg fluticasone propionate dry powder formulation equivalents total daily dose) + LABA for ≥2 months prior to enrollment (see Appendix F for medium and high daily ICS doses by formulation) 7. For patients on MD ICS/LABA, stable LTRA or LAMA (≥2 weeks) is allowed 8. Documented at least one exacerbation in the year prior to enrolment
* A qualifying historical asthma exacerbation is a symptomatic worsening requiring systemic corticosteroid (i.e., oral, intravenous (IV) or intramuscular; any healthcare setting or temporary increase from a stable maintenance dose of oral corticosteroid) or that resulted in hospitalization or emergency room/urgent care visit.

  * Source documentation is required for physician-diagnosed asthma, ICS-LABA use and asthma exacerbations over the prior year. A patient verbal history suggestive of asthma symptoms and/or prior asthma exacerbations, but without supporting documentation, is not sufficient to satisfy these inclusion criteria.
  * Examples of acceptable documentation of the asthma disease state and prior asthma exacerbations include clinic visit (primary or specialist Health care provider (HCP)), emergency room/urgent care, or hospital records listing asthma as a current problem, plus documentation of at least 1 asthma exacerbations during the 12 months prior to ICF.

Weight 9. Weight of ≥40 kg. Sex and Contraceptive/Barrier Requirements 10. Male and/or female Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

* Female patients:
* Females not of childbearing potential are defined as females who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Females will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to Visit 1(Week -1 to Week 0) without an alternative medical cause. The following age-specific requirements apply:
* Females < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and FSH levels in the postmenopausal range.
* Females ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.
* Female patients of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Females of childbearing potential who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control, as defined below, from enrolment throughout the study and until at least 12 weeks after last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician.
* The following are not acceptable methods of contraception: periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea. Female condom and male condom should not be used together.
* All WOCBP must have a negative serum pregnancy test result at Visit 1(Week -1 to Week 0).
* Highly effective birth control methods include: Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the patient (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments) [(periodic abstinence eg, calendar, ovulation,symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to study intervention, and withdrawal are not acceptable methods of contraception], a vasectomised partner, Implanon®, bilateral tubal occlusion, intrauterine device/levonorgestrel intrauterine system, Depo-Provera™ injections, oral contraceptive, and Evra Patch™, Xulane™, or NuvaRing®.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the potential for benralizumab treated patients to reduce their standard of care asthma controller regimen in the overall patient population and by subgroups of baseline background therapy Subgroups of background therapy | within 40 weeks after the first administration
  Main outcomes: Proportion of patients with at least one controller medication category reduction at end of reduction phase
  * discontinuation of LTRA, or
  * discontinuation of LAMA, or
  * getting to MD ICS/LABA or
  * getting to LD ICS/LABA

SECONDARY OUTCOMES:
To assess standard asthma efficacy measures for benralizumab treated patients when reducing their standard of care asthma controller regimen for pulmonary function measured by pre-BD FEV1 | From 16~40 weeks
  Change in pre-BD FEV1 measured in litres from beginning of reduction phase to end of reduction phase & FEV1 < -100mL compared to beginning of reduction phase
To assess standard asthma efficacy measures for benralizumab treated patients when reducing their standard of care asthma controller regimen for asthma symptoms control measured by ACQ-5 & SGRQ Score | From 16~40 weeks
  * Change in measured by ACQ-5 score & SGRQ score from beginning of reduction phase to end of reduction phase
  * Measured by Proportion of patients with no deterioration (defined as ACQ-5 score change <0.5 score since last visit) during reduction phase
To assess standard asthma efficacy measures for benralizumab treated patients at induction phase in the overall patient population and by subgroups of baseline background therapy | from 0-16 weeks
  * Change in FEV1 in litres from beginning of induction phase to end of induction phase
  * Change in ACQ-5 score and SGRQ score from beginning of induction phase to end of induction phase
  * Proportion of patients achieving ACQ-5 MCID improvement (defined as change in ACQ-5 score≤-0.5 score compared to beginning of induction phase) and SGRQ MCID improvement (defined as change in SGRQ score ≤-4 score compared to beginning of induction phase) during induction phase
To assess standard asthma efficacy measures for benralizumab treated patients at induction phase in the overall patient population and by subgroups of baseline background therapy | within 0-16 weeks after first administration
  * Change in measured by ACQ-IA score from beginning of induction phase to end of induction phase
  * Measured by Proportion of patients achieving ACQ-IA score MCID improvement (defined as change in ACQ-IA score ≤-0.5 compared to beginning of induction phase) at end of induction phase
To assess overall asthma exacerbation rate during the study of severe eosinophilic asthma patients treated with benralizumab in the overall patient population and by subgroups of baseline background therapy | within 56 weeks after first administration
  * Annualized asthma exacerbation rate during the study (from first dose to EOT) and 1-year baseline period
  * Change in annualized asthma exacerbation rate during study phase vs. 1-year baseline period
  Annualized asthma exacerbation rate Defined as Number of exacerbations×365.25/(Follow-Up Date-First Benralizumab dose date+1)
To assess biomarkers of severe eosinophilic asthma patients treated with benralizumab in the overall patient population and by subgroups of baseline background therapy | from -1 week to 60 week
  Baseline and follow-up visits, and change from baseline:
  Blood EOS measured as cells per litre
To assess biomarkers of severe eosinophilic asthma patients treated with benralizumab in the overall patient population and by subgroups of baseline background therapy | from -1 week to 56 week
  Baseline and follow-up visits, and change from baseline:· FeNO measured as parts per billion
To assess the safety and tolerability of benralizumab during the study in patients with severe eosinophilic asthma, while reducing their standard of care asthma controller regimen and maintaining asthma symptom control. | from -1 week to 60 week
  * Frequency of Adverse Events/Serious Adverse Events
  * Vital Signsa
  * Laboratory variables (chemistry and hematology)
To assess biomarkers of severe eosinophilic asthma patients treated with benralizumab in the overall patient population and by subgroups of baseline background therapy | from -1 week to 56 week
  Baseline and follow-up visits, and change from baseline:· IgE measured as per

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhang, Professor, Principal Investigator — ShangHai First General Hospital; HuaHao Shen, Professor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (38):
- China (38):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huzhou
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Luoyang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tangshan
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuhu
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhangzhou
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/